CLINICAL TRIAL: NCT02058823
Title: Cardiovascular and Metabolic Physiological Adaptations to Intermittent Hypoxia. Physiological Aspects and Expression of Receptors and Cellular Mediators
Brief Title: Intermittent Hypoxia 2: Cardiovascular and Metabolism
Acronym: IH2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: budget constraints
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2011-32; P-2011-32-HI2 (Other: CPP Caen)
Record Dates: First submitted 2012-04-18; First posted 2014-02-10 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Hypoxia; Sleep Apnea; Obstructive Sleep Apnea
Keywords: Hypoxia; Sleep apnea; Valsartan; Amlodipine; Healthy subjects; Randomized; Cross-over; International; Sympathetic nervous system
MeSH Terms: conditions — Hypoxia; Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Valsartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: Real hypoxia and ¨Placebo (Placebo Comparator): This arm last 4 weeks with 2 periods of 2 weeks separated by a 6 weeks wash-out. The subjects of this arm receive the real hypoxia and the placebo during the first two weeks and, after the wash-out, receive the treatment of the arm 2.
  Interventions: Drug: Placebo
- Arm 2: Hypoxia placebo and Placebo (Placebo Comparator): This arm last 4 weeks with 2 periods of 2 weeks separated by a 6 weeks wash-out. The subjects of this arm receive the hypoxia placebo and the placebo during the first two weeks and, after the wash-out, receive the treatment of the arm 1.
  Interventions: Drug: Placebo
- Arm 3: Hypoxia and Valsartan (Active Comparator): This arm last 4 weeks with 2 periods of 2 weeks separated by a 6 weeks wash-out. The subjects of this arm receive the real hypoxia and the Valsartan during the first two weeks and, after the wash-out, receive the treatment of the arm 4.
  Interventions: Drug: Valsartan
- Arm 4: Hypoxia and Amlodipine (Active Comparator): This arm last 4 weeks with 2 periods of 2 weeks separated by a 6 weeks wash-out. The subjects of this arm receive the real hypoxia and the amlodipine during the first two weeks and, after the wash-out, receive the treatment of the arm 3.
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Placebo — The subjects receive 1 oral pill of placebo each morning during the second week of the two periods, so 14 pills in all.
  Other Names: Placebo Valsartan
  Arms: Arm 1: Real hypoxia and ¨Placebo
Drug: Placebo — The subjects receive 1 oral pill of placebo each morning during the second week of the two periods, so 14 pills in all.
  Other Names: Placebo Almodipine
  Arms: Arm 2: Hypoxia placebo and Placebo
Drug: Valsartan — The subjects receive 1 oral pill of Valsartan each morning during the second week of the two periods, so 14 pills in all. 1 pill equal 40 mg.
  Other Names: Tareg
  Arms: Arm 3: Hypoxia and Valsartan
Drug: Amlodipine — The subjects receive 1 oral pill of Amlodipine each morning during the second week of the two periods, so 14 pills in all. 1 pill equal 6,944 mg of amlodipine besilate with 5 mg of amlodipine.
  Other Names: Effective Amlodipine
  Arms: Arm 4: Hypoxia and Amlodipine

SUMMARY:
The purpose of this study is to compare cardiovascular physiological adaptation to intermittent hypoxia (IH) of nonobese healthy subjects. The exposure will be two periods of two weeks (IH versus exposure "placebo hypoxia"). The investigators will use pharmacological tools, peripheral vasodilator (amlodipine) or specific blocker of angiotensin receptor (valsartan) versus the taking of a placebo. The allocation of the tool and the exhibition will be randomized (HI / placebo, valsartan / amlodipine). The outcome measures evaluated concern the cardiovascular system, systemic inflammation and tissular and glucose metabolism.

The investigators assume an increase in arterial resistance during the intermittent hypoxia compared to the control group, these being dependent on sympathetic tone.

The investigators hypothesize that the metabolic alterations that will be observed after experimental simulation (IH and fragmentation of sleep for 15 consecutive nights) will be less severe in the valsartan group than in the amlodipine group in comparison with the placebo group.

A serum bank and a gene bank will be performed for the requirements of subsequent studies if necessary.

DETAILED DESCRIPTION:
There are many physiological situations in which the organism is exposed to hypoxia, such as exercise and altitude. In addition some pathological situations also involve hypoxia, such as obesity, heart failure, respiratory failure and sleep apnea syndrome.

Hypoxia associated with altitude is frequently marked by the presence of sleep during periodic breathing induces a particular pattern of hypoxia called intermittent hypoxia. Also some subjects are "intolerant altitude" and develop specific pathologies at high altitude (acute mountain evil, pulmonary edema ...).

We recently demonstrated that subjects tolerate the altitude had just intermittent hypoxia while they were sleeping during the simulated altitude. The protective role of intermittent hypoxia in the mechanisms of occurrence of intolerance to altitude remains to be understood more precisely. In fact those who were intolerant to altitude has no periodic breathing and therefore intermittent hypoxia during the oxygen-deficient atmosphere.

Conversely, the sleep apnea syndrome (SAS) also characterized by a HI. It is produced by repeated episodes of airway obstruction during sleep, producing a sequence: respiratory effort, hypoxia / re-oxygenation and sleep interruption.

The HI is associated with both a well established cardiovascular morbidity but also to cardioprotection. This relates to cardiovascular morbidity rise in blood pressure can certainly promote the development after many years of hypertension. On the other hand the presence of sleep apnea syndrome is advanced as a factor favoring the coronary collateral circulation and therefore will bring a cardioprotective effect for patients.

Understanding the mechanisms of physiological adaptations to intermittent hypoxia by passing a deleterious evolution of a protective HI is therefore critical.

Exposure to altitude or OSAS induces the activation of intermediary mechanisms such as sympathetic activation, altered vascular reactivity, systemic inflammation and low-grade oxidative stress. The direct involvement of these mechanisms is dependent mainly intermediate of intermittent hypoxia. The shift in equilibrium between activator and inhibitor factors will evolve either to a protective mode (adaptation to altitude) or pathologic (cardiovascular complication of OSA).

Sympathetic activation has been demonstrated in patients with OSAS, reversible with effective treatment. The importance of cardiovascular sympathetic activation in elevating blood pressure by intermittent hypoxia is shown in animal models of HI. We also found an increase in sympathetic activation in our reversible model of HI in healthy subjects.

The elevation of that sympathetic activity is assumed to be multifactorial. An increase in tone but also a central potentiation thereof by an increase in peripheral chemoreflex sensitivity (sensitive to hypoxia) and against a lack of regulation by the arterial baroreflex.

Moreover angiotensin system modulates the central sympathetic tone and peripheral chemoreflex sensitivity. These actions are complementary in a signaling pathway of particular interest in exposure to intermittent hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* Subject aged of 18 years-old at least
* Diagnostic AHI<15/h and <5% of total sleep time spent with a SaO2<90%
* Free and informed consent signed
* Subject covered by social security
* Negative pregnancy test

Exclusion Criteria:

* Subject with a medical pathology (respiratory, cardiovascular, renal, metabolic, neurological...)
* Tobacco consumption > 5 cigarettes/days
* Alcohol consumption > 3 units/days (1 unit=1 drink)
* Subject under trusteeship or guardianship
* Subject unaffiliated with the social security
* Person deprived of their liberty, adult protected by laws, person hospitalized
* Ongoing participation in another clinical research study
* Subject non-cooperative or respectful of obligations inherent in the participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08-07 (Actual); Primary Completion 2014-07-17 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Change in sympathetic activity | Day 1 and at Day 14
  The sympathetic activity will be directly measured by microneurography of the peroneal nerve

SECONDARY OUTCOMES:
Measure of adrenergic, inflammatory and metabolic markers in adipose tissues by chronic intermittent hypoxia versus placebo in healthy nonobese subjects. | Day 14
  The adrenergic receptors will be evaluated by immuno histochemistry appearance and by measuring mRNA levels of alpha and beta and AT1 and AT2 receptors by RT-PCR on total RNA extracted from the subcutaneous adipose tissue.
  Insulin sensitivity test would be performed on adipose tissues.
Measure variations in parameters of inflammation in adipose tissue by chronic intermittent hypoxia versus placebo in healthy nonobese subjects. | Day 14
  The inflammation will be assessed by measuring mRNA levels of proinflammatory cytokines and anti-inflammatory (IL-1, IL-6, IL-4, IL-10, IL-12, RANTES, TNF, leptin, adiponectin, CD68 (macrophage inflammation)) by RT-PCR on total RNA extracted (Mirvana, Ambion) from the subcutaneous adipose tissue.
Measure of metabolic aspects of the OGTT test. | Day 14
  Measure of glucose intolerance and insulin sensitivity inducing by intermittent hypoxia by multisamples OGTT test.
Measure the activation of systemic inflammation by chronic HI versus placebo in healthy nonobese subjects. The systemic inflammation will be assessed in non-stress and during the OGTT. | Day 14
  * Non-stress: by measuring the cytokines pro-and anti-inflammatory (IL-1, IL-6, IL-4, IL-10, IL-12, RANTES, TNF, leptin, adiponectin, CD68).
  * OGTT: Kinetics concentrations of C-reactive protein, TNF-α, IL6, IL8, IL1-ß, CCL2/MCP-1, PAI-1, IL-1 Ra, IL-10.
Assessing markers implicated in the pathophysiology of chronic metabolic diseases after HI versus placebo in healthy nonobese subjects during OGTT. | Day 14
  * Psychology:Hunger, appetite and food preference by validated questionnaires.
  * Behavior:Calorie intake, food choices, energy expenditure.
  * Physiology:
    * Metabolism rest:Indirect calorimetry.
    * Carbohydrate metabolism:Glucose tolerance, sensitivity to insulin, insulin secretion, time profiles of several proteins.
    * Neuroendocrine control of appetite:Temporal Patterns of hormones.
    * Lipid profiles:Temporal Patterns of FFA, concentrations of triglycerides and cholesterol.
    * Autonomic nervous system activity:Cardiac inter-beat intervals, urine sample, time profiles of catecholamines.
Change in vascular responsivness | At day 1 and Day 14
  Some others vascular beds will be explored skin, eyes before and after intermittent hypoxia.Use o f a laser doppler cutaneous, choroidal and ophthalmic arteries.
Change in Sympathetic and vascular determinant of Blood pressure | Day 1 and Day 14
  Heart rate variability and vascular flow and arterial pressure. Heart rate variability will be measure from 24h ECG recording.The vascular flow will be measured by Doppler waveform of the popliteal artery. The blood pressure will be measured by an ambulatory blood pressure monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Renaud RT Tamisier, PhD, Principal Investigator — University Hospital of Genoble
Locations (1):
- Laboratoire EFCR - Functional Cardio-respiratory Exploration Laboratory, La Tronche, Isère, France

REFERENCES:
- [Background] Steiner S, Schueller PO, Schulze V, Strauer BE. Occurrence of coronary collateral vessels in patients with sleep apnea and total coronary occlusion. Chest. 2010 Mar;137(3):516-20. doi: 10.1378/chest.09-1136. Epub 2009 Oct 26. PMID 19858231
- [Background] Lavie L. Obstructive sleep apnoea syndrome--an oxidative stress disorder. Sleep Med Rev. 2003 Feb;7(1):35-51. doi: 10.1053/smrv.2002.0261. PMID 12586529
- [Background] Shamsuzzaman AS, Gersh BJ, Somers VK. Obstructive sleep apnea: implications for cardiac and vascular disease. JAMA. 2003 Oct 8;290(14):1906-14. doi: 10.1001/jama.290.14.1906. PMID 14532320
- [Background] Carlson JT, Hedner J, Elam M, Ejnell H, Sellgren J, Wallin BG. Augmented resting sympathetic activity in awake patients with obstructive sleep apnea. Chest. 1993 Jun;103(6):1763-8. doi: 10.1378/chest.103.6.1763. PMID 8404098
- [Background] Somers VK, Dyken ME, Clary MP, Abboud FM. Sympathetic neural mechanisms in obstructive sleep apnea. J Clin Invest. 1995 Oct;96(4):1897-904. doi: 10.1172/JCI118235. PMID 7560081
- [Background] Hedner J, Darpo B, Ejnell H, Carlson J, Caidahl K. Reduction in sympathetic activity after long-term CPAP treatment in sleep apnoea: cardiovascular implications. Eur Respir J. 1995 Feb;8(2):222-9. doi: 10.1183/09031936.95.08020222. PMID 7758555
- [Background] Fletcher EC, Lesske J, Culman J, Miller CC, Unger T. Sympathetic denervation blocks blood pressure elevation in episodic hypoxia. Hypertension. 1992 Nov;20(5):612-9. doi: 10.1161/01.hyp.20.5.612. PMID 1428112
- [Background] Tamisier R, Pepin JL, Remy J, Baguet JP, Taylor JA, Weiss JW, Levy P. 14 nights of intermittent hypoxia elevate daytime blood pressure and sympathetic activity in healthy humans. Eur Respir J. 2011 Jan;37(1):119-28. doi: 10.1183/09031936.00204209. Epub 2010 Jun 4. PMID 20525723
- [Background] Narkiewicz K, van de Borne PJ, Montano N, Dyken ME, Phillips BG, Somers VK. Contribution of tonic chemoreflex activation to sympathetic activity and blood pressure in patients with obstructive sleep apnea. Circulation. 1998 Mar 17;97(10):943-5. doi: 10.1161/01.cir.97.10.943. PMID 9529260
- [Background] Carlson JT, Hedner JA, Sellgren J, Elam M, Wallin BG. Depressed baroreflex sensitivity in patients with obstructive sleep apnea. Am J Respir Crit Care Med. 1996 Nov;154(5):1490-6. doi: 10.1164/ajrccm.154.5.8912770.
- [Background] Punjabi NM, Beamer BA. Alterations in Glucose Disposal in Sleep-disordered Breathing. Am J Respir Crit Care Med. 2009 Feb 1;179(3):235-40. doi: 10.1164/rccm.200809-1392OC. Epub 2008 Nov 14. PMID 19011148
- [Background] Spiegel K, Tasali E, Leproult R, Van Cauter E. Effects of poor and short sleep on glucose metabolism and obesity risk. Nat Rev Endocrinol. 2009 May;5(5):253-61. doi: 10.1038/nrendo.2009.23. PMID 19444258
- [Background] Larsen JJ, Hansen JM, Olsen NV, Galbo H, Dela F. The effect of altitude hypoxia on glucose homeostasis in men. J Physiol. 1997 Oct 1;504 ( Pt 1)(Pt 1):241-9. doi: 10.1111/j.1469-7793.1997.241bf.x. PMID 9350634
- [Background] Braun B, Rock PB, Zamudio S, Wolfel GE, Mazzeo RS, Muza SR, Fulco CS, Moore LG, Butterfield GE. Women at altitude: short-term exposure to hypoxia and/or alpha(1)-adrenergic blockade reduces insulin sensitivity. J Appl Physiol (1985). 2001 Aug;91(2):623-31. doi: 10.1152/jappl.2001.91.2.623. PMID 11457773
- [Background] Spiegel K, Knutson K, Leproult R, Tasali E, Van Cauter E. Sleep loss: a novel risk factor for insulin resistance and Type 2 diabetes. J Appl Physiol (1985). 2005 Nov;99(5):2008-19. doi: 10.1152/japplphysiol.00660.2005. PMID 16227462
- [Background] Spiegel K, Leproult R, Colecchia EF, L'Hermite-Baleriaux M, Nie Z, Copinschi G, Van Cauter E. Adaptation of the 24-h growth hormone profile to a state of sleep debt. Am J Physiol Regul Integr Comp Physiol. 2000 Sep;279(3):R874-83. doi: 10.1152/ajpregu.2000.279.3.R874. PMID 10956244
- [Background] Spiegel K, Leproult R, L'hermite-Baleriaux M, Copinschi G, Penev PD, Van Cauter E. Leptin levels are dependent on sleep duration: relationships with sympathovagal balance, carbohydrate regulation, cortisol, and thyrotropin. J Clin Endocrinol Metab. 2004 Nov;89(11):5762-71. doi: 10.1210/jc.2004-1003. PMID 15531540
- [Background] Spiegel K, Leproult R, Van Cauter E. Impact of sleep debt on metabolic and endocrine function. Lancet. 1999 Oct 23;354(9188):1435-9. doi: 10.1016/S0140-6736(99)01376-8. PMID 10543671
- [Background] Tamisier R, Gilmartin GS, Launois SH, Pepin JL, Nespoulet H, Thomas R, Levy P, Weiss JW. A new model of chronic intermittent hypoxia in humans: effect on ventilation, sleep, and blood pressure. J Appl Physiol (1985). 2009 Jul;107(1):17-24. doi: 10.1152/japplphysiol.91165.2008. Epub 2009 Feb 19. PMID 19228987
- [Background] Gilmartin GS, Lynch M, Tamisier R, Weiss JW. Chronic intermittent hypoxia in humans during 28 nights results in blood pressure elevation and increased muscle sympathetic nerve activity. Am J Physiol Heart Circ Physiol. 2010 Sep;299(3):H925-31. doi: 10.1152/ajpheart.00253.2009. Epub 2010 Jun 25. PMID 20581089
- [Background] Bilo G, Caldara G, Styczkiewicz K, Revera M, Lombardi C, Giglio A, Zambon A, Corrao G, Faini A, Valentini M, Mancia G, Parati G. Effects of selective and nonselective beta-blockade on 24-h ambulatory blood pressure under hypobaric hypoxia at altitude. J Hypertens. 2011 Feb;29(2):380-7. doi: 10.1097/HJH.0b013e3283409014. PMID 21045724
- [Background] Gilmartin GS, Tamisier R, Curley M, Weiss JW. Ventilatory, hemodynamic, sympathetic nervous system, and vascular reactivity changes after recurrent nocturnal sustained hypoxia in humans. Am J Physiol Heart Circ Physiol. 2008 Aug;295(2):H778-85. doi: 10.1152/ajpheart.00653.2007. Epub 2008 Jun 6. PMID 18539753
- [Background] Tamisier R, Anand A, Nieto LM, Cunnington D, Weiss JW. Arterial pressure and muscle sympathetic nerve activity are increased after two hours of sustained but not cyclic hypoxia in healthy humans. J Appl Physiol (1985). 2005 Jan;98(1):343-9. doi: 10.1152/japplphysiol.00495.2004. Epub 2004 Sep 24. PMID 15448121
- [Background] Tamisier R, Hunt BE, Gilmartin GS, Curley M, Anand A, Weiss JW. Hemodynamics and muscle sympathetic nerve activity after 8 h of sustained hypoxia in healthy humans. Am J Physiol Heart Circ Physiol. 2007 Nov;293(5):H3027-35. doi: 10.1152/ajpheart.00277.2007. Epub 2007 Sep 14. PMID 17873026
- [Background] Tamisier R, Nieto L, Anand A, Cunnington D, Weiss JW. Sustained muscle sympathetic activity after hypercapnic but not hypocapnic hypoxia in normal humans. Respir Physiol Neurobiol. 2004 Jul 20;141(2):145-55. doi: 10.1016/j.resp.2004.04.006. PMID 15239965
- [Background] Garet M, Barthelemy JC, Degache F, Pichot V, Duverney D, Roche F. Modulations of human autonomic function induced by positive pressure-assisted breathing. Clin Physiol Funct Imaging. 2006 Jan;26(1):15-20. doi: 10.1111/j.1475-097X.2005.00645.x. PMID 16398665
- [Background] Roche F, Barthelemy JC, Garet M, Duverney D, Pichot V, Sforza E. Continuous positive airway pressure treatment improves the QT rate dependence adaptation of obstructive sleep apnea patients. Pacing Clin Electrophysiol. 2005 Aug;28(8):819-25. doi: 10.1111/j.1540-8159.2005.00188.x. PMID 16105010
- [Background] Roche F, Gaspoz JM, Court-Fortune I, Minini P, Pichot V, Duverney D, Costes F, Lacour JR, Barthelemy JC. Screening of obstructive sleep apnea syndrome by heart rate variability analysis. Circulation. 1999 Sep 28;100(13):1411-5. doi: 10.1161/01.cir.100.13.1411. PMID 10500042
- [Background] Spiegel K, Tasali E, Penev P, Van Cauter E. Brief communication: Sleep curtailment in healthy young men is associated with decreased leptin levels, elevated ghrelin levels, and increased hunger and appetite. Ann Intern Med. 2004 Dec 7;141(11):846-50. doi: 10.7326/0003-4819-141-11-200412070-00008. PMID 15583226
- [Background] Tasali E, Leproult R, Ehrmann DA, Van Cauter E. Slow-wave sleep and the risk of type 2 diabetes in humans. Proc Natl Acad Sci U S A. 2008 Jan 22;105(3):1044-9. doi: 10.1073/pnas.0706446105. Epub 2008 Jan 2. PMID 18172212
- [Background] Hoppeler H, Vogt M. Hypoxia training for sea-level performance. Training high-living low. Adv Exp Med Biol. 2001;502:61-73. doi: 10.1007/978-1-4757-3401-0_6. PMID 11950155
- [Background] Somers VK, White DP, Amin R, Abraham WT, Costa F, Culebras A, Daniels S, Floras JS, Hunt CE, Olson LJ, Pickering TG, Russell R, Woo M, Young T; American Heart Association Council for High Blood Pressure Research Professional Education Committee, Council on Clinical Cardiology; American Heart Association Stroke Council; American Heart Association Council on Cardiovascular Nursing; American College of Cardiology Foundation. Sleep apnea and cardiovascular disease: an American Heart Association/american College Of Cardiology Foundation Scientific Statement from the American Heart Association Council for High Blood Pressure Research Professional Education Committee, Council on Clinical Cardiology, Stroke Council, and Council On Cardiovascular Nursing. In collaboration with the National Heart, Lung, and Blood Institute National Center on Sleep Disorders Research (National Institutes of Health). Circulation. 2008 Sep 2;118(10):1080-111. doi: 10.1161/CIRCULATIONAHA.107.189375. Epub 2008 Aug 25. No abstract available. PMID 18725495